CLINICAL TRIAL: NCT04268212
Title: Effects of Bitter Melon Intake and Moderate-Intensity Physical Activity on Postprandial Glucose Responses in Type 2 Diabetic Patients
Brief Title: An Alternative Approach to Improve Hyperglycemia Among Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004172
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bitter Melon (Experimental): The participants were asked to consume 100 ml of bitter melon juice 15 minutes prior to the 75-g oral glucose intake. Participants drank the juice within 5 minutes. Participants remained seated throughout the following 2 hours.
  Interventions: Dietary Supplement: Bitter melon juice (100 ml)
- Exercise (Experimental): Participants performed 30 minutes of treadmill walking at 65% of the age-predicted maximum heart rate. The exercise started 15 minutes after the 75-g oral glucose intake.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: Bitter melon juice (100 ml) — Fresh bitter melon fruits were purchased from certified local groceries. The seeds of bitter melon were removed, and the juice was obtained from the raw fruit using a blender. Every 140 g of bitter melon fruit produced approximately 100 ml bitter melon juice.
  Arms: Bitter Melon
Behavioral: Exercise — The walking exercise was started 15 minutes after the glucose load. Walking speed was determined to elicit 65% of the maximum heart rate (HRmax) during exercise for each participant. HRmax was estimated using the America College of Cardiology prediction model, HRmax=208 - 0.7 × age. All participants wore a heart rate monitor (Polar, Vantage, XL) around the chest to assess exercise intensity. A rate of perceived exertion was assessed every 2 minutes based on the Borg's scale.
  Arms: Exercise

SUMMARY:
The study compared the effect of bitter melon intake and moderate exercise on postprandial glucose levels as measured by incremental area under the curve (iAUC) in eight patients with type 2 diabetes.

DETAILED DESCRIPTION:
Background: This study compared the effects of bitter melon intake and moderate-intensity physical activity on postprandial glucose responses in type 2 diabetic patients.

Methods: A total of 8 patients with type 2 diabetes were randomly assigned to two sequences (AB, BA) with two treatments (A or B) using a 2 x 2 randomized cross-over design: A) 100 ml of bitter melon juice administered 15 minutes prior to the 75-g oral glucose load; B) 30 minutes walking at moderate-intensity performed 15 minutes after the oral glucose load.

ELIGIBILITY:
Inclusion Criteria:

* An age of 20 to 79 years
* Physician-diagnosed type 2 diabetes
* Medical clearance for physical activity from their healthcare provider

Exclusion Criteria:

* Pregnant or were receiving insulin treatment
* An allergy to bitter melon
* Medical conditions that impacted the normal the functioning of the gastrointestinal tract
* Contraindications to physical activity

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-09-20 (Actual)

PRIMARY OUTCOMES:
mean glucose | 2-hour postprandial period
  mean glucose values
incremental area under the curve | 2-hour postprandial period
  2-hour postprandial glucose incremental area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lee, Ph.D., Principal Investigator — Arizona State University

IPD SHARING:
Plan to Share IPD: No